CLINICAL TRIAL: NCT01243658
Title: "The Effects of Oxytocin on Patients With Borderline Personality Disorder"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Markus Heinrichs (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Markus Heinrichs, Prof. Dr. Markus Heinrichs, University of Freiburg
Organization: University of Freiburg (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: OX02
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Effects of Oxytocin on Borderline Personality Disorder; Borderline Personality Disorder
Keywords: Oxytocin; BPD; Borderline
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxytocin (Experimental): Oxytocin
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Oxytocin — Oxytocin
  Arms: Oxytocin
Other: placebo — placebo
  Arms: Placebo

SUMMARY:
RCT. Two substudies (clinical and experimental). Main objective of the trial is to examine if oxytocin, compared to placebo shows any additional effect on the therapy achievements (outcome) of patients with borderline personality disorder, who receive an in-patient standard psychotherapy (Dialectical-behavioral-therapy, Marsha Linehan (2006)).

Secondary objectives :

Investigate if oxytocin compared to placebo enhances social trust and emotion recognition in patients with borderline personality disorder. Comparison of the effects of Oxytocin on patients with BPD and major depression.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Both, male and female
* Minimum Age: 18 Years
* Maximum Age: 50 Years
* Borderline personality disorder or major depression (clinical control group)
* Mini Mental Status Test > 27 (capacity to consent)

Exclusion Criteria:

* chronic or acute somatic health problems
* Schizophrenia
* Bipolar affective disorder
* pregnancy
* breast feeding
* neurological disorder
* allergy to antidegradants

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2011-01; Primary Completion 2021-04 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
BPD Symptoms | BPD Symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Markus Heinrichs, Prof. Dr., Study Director — Institut für Psychologie der Univeristät Freiburg
Locations (1):
- Albert-Ludwigs-Universität-Freiburg, Freiburg im Breisgau, Baden-Würtemberg, Germany